CLINICAL TRIAL: NCT02654912
Title: Community-led Responses for Elimination (CoRE): A Cluster Randomized Controlled Trial of Reactive Case Detection Versus Reactive Drug Administration in Malaria Elimination Areas in Southern Province Zambia
Brief Title: Community-led Responses for Elimination: Controlled Trial of Reactive Case Detection Versus Reactive Drug Administration
Acronym: CORE Zambia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Ministry of Health, Zambia (Other Government); AKROS Global Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PATH-WIRB-1155095
Record Dates: First submitted 2015-11-12; First posted 2016-01-13 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2020-09

CONDITIONS: Malaria
Keywords: malaria; elimination; surveillance and response; dihydroartemisinin+piperaquine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reactive Focal Drug Administration (Experimental): This is the experimental arm and is described by a reactive response to passively detected index case of malaria. The reactive response consists of treating all individuals within a defined radius of each RDT-confirmed incident malaria case with dihydroartemisinin-piperaquine (DHAP).
  Interventions: Drug: Reactive Focal Drug Administration
- Reactive Focal Test and Treat (No Intervention): This is the current standard of care in Southern Province and is described by a reactive response to passively detected index case of malaria. The reactive response consists of testing all individuals within a defined radius of each RDT-confirmed incident malaria case with an RDT and treating all positive individuals with artemether-lumefantrine (AL).

INTERVENTIONS:
Drug: Reactive Focal Drug Administration — This is the experimental arm and is described by a reactive response to passively detected index case of malaria. The reactive response consists of treating all individuals within a defined radius of each RDT-confirmed incident malaria case with dihydroartemisinin-piperaquine (DHAP).
  Arms: Reactive Focal Drug Administration

SUMMARY:
This study is designed to compare the effectiveness of reactive focal drug administration (RFDA) using dihydroartemisinin+piperaquine (DHAP) versus reactive focal test and treat (RFTAT) using artemether+lumefantrine (AL) as a routine process for identifying and eliminating malaria transmission as measured through achieving zero seropositivity in children under five in Southern Province, Zambia. These two strategies are potential candidates for expanded malaria operational surveillance and elimination for low malaria transmission areas.

DETAILED DESCRIPTION:
The study is a cluster randomized controlled trial designed to evaluate the impact of RFDA intervention against current standard of care for the impact on seropositivity in children under five years, passive surveillance for confirmed malaria case incidence, and elimination of transmission from hotspots. It will be conducted among a background population of ~130,000 people in ~30,000 households in 16 health center catchment areas across several districts in Southern Province. The government of Zambia is pursuing malaria elimination as a national goal on an accelerated timeline and this trial will help evaluate two treatment-based strategies for supporting malaria elimination.

The secondary objectives of the study include: 1). Compare the effectiveness of RFDA using DHAP with RFTAT using AL in reducing rapid diagnostic test (RDT) confirmed malaria incidence through passive case detection at health facilities; 2). Compare the effectiveness of RFDA using DHAP with RFTAT using AL in reducing the prevalence of malaria and preventing re-infection in individuals receiving reactive responses; 3). Compare the cost-effectiveness of RFDA using DHAP with RFTAT using AL in reducing the burden of malaria in the community; 4). Measure the proportion of P. falciparum infections likely attributable to importation and local transmission using parasite genotyping as well as defining genotype spatial distribution; 5). Assess the utility of using serology to measure short term changes in malaria transmission and evaluate malaria elimination programs; and 6). Assess the feasibility of using remotely sensed malaria risk maps to identify areas with higher potential for local malaria transmission.

ELIGIBILITY:
Inclusion Criteria:

* anyone not excluded and consenting

Exclusion Criteria:

* contraindications from manufacturer for medications including currently taking haloperidol, artane, Phenergan (Promethazine), chlorpromazine, erythromycin, Azithromycin, clarithromycin, Ketoconazole, fluconazole, mefloquine (as prophylaxis), lumefantrine (in Coartem), quinine, Septrin
* anyone seriously ill
* currently taking antimalarial medicines
* allergy to artemisinin drugs
* pregnant women in first trimester
* children under 3 months of age
* reported heart condition

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8682 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Malaria seropositivity in children under five | 24 months
  Malaria seropositivity in children under five after two-year intervention within health center catchment areas

SECONDARY OUTCOMES:
Incidence of malaria confirmed by RDT or microscopy as measured through passive case detection at health posts and health centers | 24 months
  Quality-improved incidence of malaria data confirmed by malaria rapid diagnostic test (RDT) or microscopy as measured through passive case detection at health posts and health centers in the study area.
PCR parasite prevalence among individuals participating at 0, 30 and 90 days following a reactive research response for a period of 24 months | 24 months
  Polymerase Chain Reaction (PCR)-based testing for malaria parasite prevalence of individuals participating in each community at 0, 30 and 90 days following a reactive research response for a period of 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bridges, PhD, Principal Investigator — Akros
Locations (1):
- Southern province medical office, Choma, Southern Province, Zambia

REFERENCES:
- [Background] Bridges DJ, Miller JM, Chalwe V, Moonga H, Hamainza B, Steketee R, Silumbe K, Nyangu J, Larsen DA. Community-led Responses for Elimination (CoRE): a study protocol for a community randomized controlled trial assessing the effectiveness of community-level, reactive focal drug administration for reducing Plasmodium falciparum infection prevalence and incidence in Southern Province, Zambia. Trials. 2017 Nov 2;18(1):511. doi: 10.1186/s13063-017-2249-0. PMID 29096671
- [Derived] Bridges DJ, Miller JM, Chalwe V, Moonga H, Hamainza B, Steketee RW, Mambwe B, Mulube C, Wu L, Tetteh KKA, Drakeley C, Chishimba S, Mwenda M, Silumbe K, Larsen DA. Reactive focal drug administration associated with decreased malaria transmission in an elimination setting: Serological evidence from the cluster-randomized CoRE study. PLOS Glob Public Health. 2022 Dec 5;2(12):e0001295. doi: 10.1371/journal.pgph.0001295. eCollection 2022. PMID 36962857